CLINICAL TRIAL: NCT02504307
Title: Randomized Evaluation of Vascular Healing After Implantation of Sirolimus Eluting Stent Inspiron™ Versus Its Own Bare Metal Version- An OCT Evaluation After 3 Months Follow-up
Brief Title: OCT Evaluation 3 Months After Sirolimus Eluting Stent Implantation
Acronym: Laranjeiras
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Scitech Produtos Medicos Ltda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Laranjeiras
Record Dates: First submitted 2015-07-20; First posted 2015-07-21 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inspiron (Experimental): Sirolimus Eluting Stent Inspiron
  Interventions: Device: Sirolimus Eluting Stent Inspiron
- Cronus (Active Comparator): Bare Metal Stent
  Interventions: Device: Bare Metal Stent

INTERVENTIONS:
Device: Sirolimus Eluting Stent Inspiron — Angioplasty with Sirolimus Eluting Stent Inspiron implantation
  Arms: Inspiron
Device: Bare Metal Stent — Angioplasty with Bare Metal Stent Cronus implantation
  Arms: Cronus

SUMMARY:
Prospective, single center, randomized and non-inferiority study, to include up to 60 patients with de novo coronary artery disease. Patients will be followed at 30 days, 3, 6 and 12 months. At 3 months all patients will be submitted to angiographic and OCT evaluation.

ELIGIBILITY:
Inclusion Criteria:

* one or two de novo lesions (> 50% visual estimation)
* lesion diameter between 2.5 and 3.5 mm
* lesion length up to 33 mm.

Exclusion Criteria:

* MI within the last 72 hours
* restenotic lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-07; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Safety | 3 months
  Percentage of strut coverage by OCT

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Leandro, MD, Principal Investigator — Insituto Nacional de Cardiologia
Locations (1):
- Instituto Nacional de Cardiologia, Rio de Janeiro, Rio de Janeiro, Brazil